CLINICAL TRIAL: NCT06417333
Title: A Smart-wrist Band Connected Mobile Application for the Assessment and Management of Dementia Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Baris Ceyhan, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 230086
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dementia, Mild
Keywords: dementia health data fitness tracking
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: 2 15 people groups were distributes wristbands during a 6 month span
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: xiaomi mi band 7 smart wristband — Patients with mild dementia have been distributed xiaomi mi band 7 smart wristbands for health data collection

SUMMARY:
In this study, we developed a mobile application that will enable caregivers to continuously monitor the vital health, medication, activity, and location of the patients with MCI with a smart wristband while enabling them caregivers to track the progress of the disease by a machine learning model that predicts MMSE of the patient using speech

DETAILED DESCRIPTION:
3-month vital health data collection has been performed on 30 participants who are over 60 years old via smart fitness wristbands distributed to them. A mobile application has been developed that caregivers can register their patients, wristbands and allow them to monitor their health data along with their location. medication and activities while synchronizing data anonymously to the application database.

The data collection has been performed with relatively cheap, simple Xiaomi MI Band 7 wristbands that track only HR, RHR, sleep, steps and move minutes due to reasonable price and light weight and easy wearability of these devices.

Mobile application synchronizes data from wristband to application servers continuously using Google Fit services that synchronize with device software. This made it possible for the patient's data to still be collected when he or she is not using any of them.

MMSE scores of patients were taken at the beginning and at the end of the 3 month period to correlate scores with the collected aggregated health data and patient information

ELIGIBILITY:
Inclusion Criteria:

* Older patients who are willing to wear a smart wristband and have an Android smart phone

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Each participant's written Mini Mental State Examination (MMSE) score was taken in the first and last week of data collection period | 3 months
  The Mini Mental State Examination (MMSE) is a tool that can be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30, minimum is 0. A score of 24 or lower is indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Suzek, Dr., Study Chair — Head of The Bioinformatics Department
Locations (1):
- Mugla Sitki Kocman University - Dementia Clinic, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No